CLINICAL TRIAL: NCT02281812
Title: Impact of Radiofrequency Ablation on Surgical Margins in Early Stage of Malignant Breast Tumors
Brief Title: Radiofrequency Ablation in Breast Cancer
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Increased local adverse effect (breast inflamation and infection)
Sponsor: Hospital Universitari de Bellvitge (Other)
Responsible Party: Principal Investigator, Amparo Garcia-Tejedor, MD PhD, Hospital Universitari de Bellvitge
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: AC133/12
Record Dates: First submitted 2014-10-30; First posted 2014-11-04 (Estimated); Last update posted 2018-06-04 (Actual); Status verified 2018-05

CONDITIONS: Breast Cancer
Keywords: Ablation Technique; Breast cancer; Stage 1; Lumpectomy
MeSH Terms: conditions — Breast Neoplasms | interventions — Radiofrequency Ablation

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (2):
- RFA group (Experimental): A percutaneous (utlrasound-guided) radiofrequency ablation (RFA) of the tumor will be performed by the radiologist under general anesthesia. Immediately after, excision of the tumor with appropriate margin will be accomplished.
  Interventions: Procedure: Radiofrequency ablation
- Control group (No Intervention): Normal excision of the tumor according to the protocol

INTERVENTIONS:
Procedure: Radiofrequency ablation — After tumor ablation and excision of the tumor, the pathologist performed a macroscopic study of the specimen,measuring the distance between the tumor and the margin in order to indicate if extensions are mandatory. Secondly and delayed, margins will be evaluated microscopically by H&E stain. Furthermore, the tumoral viability in the ablation zone will be evaluated by NADH-diaphorase, COX and tunnel.
  Arms: RFA group

SUMMARY:
Background/Main objective: Radiofrequency ablation (RFA) is a minimally invasive procedure widespread accepted in the treatment of different tumors, especially in the liver but its benefit is not yet well-known in breast cancer.

Our main objective is to evaluate the usefulness of RFA in < 2cm malignant breast tumors to reduce the proportion of positive margins.

Methodology: The investigator propose a single-center, single-blind, phase I and II randomized controlled trial. Phase I:Security of the cool-tip cluster electrode assessing the potential adverse effects in three stages: initial,intermediate and final. Phase II: Randomized clinical trial, 2 parallel groups with 37 patients in each one.

Experimental group: percutaneous RFA previous to conventional lumpectomy. Control group: conventional surgery with lumpectomy. The number of positive margins in both groups, and the need of extending margin resection will be assessed intraoperatively. Inclusion criteria: women >40 years, infiltrating ductal breast carcinoma by biopsy. The tumor must be unique, visible by ultrasound, smaller than 2cm and located > 1 cm from the chest wall and the skin. Patients will be followed up for a period of two years to assess cosmetic result, short -term and long -term complications and recurrences.

Expected results: The "cool-tip" (cluster) ablation method reduces by at least 30% the risk of intraoperative extensions for positive margins during lumpectomy compared to conventional surgery in breast tumors with a diameter < 2 cm.

Therefore this procedure may reduce the risk of second surgeries and the removed volume of tissue.Consequently the final cosmetic result should be improved.

DETAILED DESCRIPTION:
Main objectives of the project:

* To evaluate the usefulness of radiofrequency ablation (RFA) to achieve a lower percentage of positive margins.
* To validate clinically the efficacy and safety of the method in breast tumors smaller than < 2 cm.

Specific objectives of the project:

1. To demonstrate that , after RFA, clear margins are increased in the intraoperative pathological analysis compared to conventional surgery.

   1. To quantify the number of positive margins requiring intraoperative extension in each patient, comparing the ratio in both groups.
   2. To quantify the percentage of patients requiring intraoperative extension compared in both groups.
2. To demonstrate a reduction in the volume of breast tissue removed after RFA compared to conventional surgery.

   1. Comparing in both groups the anteroposterior, transverse and craniocaudal diameters of the excised specimen, measured in cm, and to calculate the volume.
   2. Tumor weight in grams (including extensions) will be measured to compare the weights in both groups.
3. To evaluate the differences in cosmetic outcome after RFA versus conventional surgery.

   a. An international scale will be used and the scores will be compared. There will be two independent assessments, one for the physician and another for the patient.
4. To demonstrate the effectiveness of the RFA by cluster "cool-tip" electrode in the experimental group.

   1. RFA is considered as complete when no viable tumor tissue is evidenced by oxidation-reduction reaction mediated by NADH-diaphorase after surgical resection. Mitochondrial dysfunction will be also evaluated by semiquantitative and quantitative method using the enzyme cytochrome c oxidase or Complex IV (COX) and tunel. Any residual viable tumor tissue will be considered as incomplete RFA.
   2. Risk factors for incomplete ablations will be analyzed, especially tumor vascularization.
5. To demonstrate the safety of RFA by cluster "cool-tip" electrode in breast cancer tumors a. To quantify all side effects that may occur after the RFA and / or surgery and to correlate the complication rate in each group with severity.

ELIGIBILITY:
Inclusion Criteria:

* Breast single tumor,
* Clearly visible by ultrasound,
* Diameter < 2 cm
* Located >1 cm from the chest wall and skin;
* Ductal carcinoma according to previous biopsy,
* < 20% of intraductal carcinoma

Exclusion Criteria:

* Breast cancer in men;
* Personal history of ipsilateral breast cancer;
* Age <40 years;
* Pregnancy or breastfeeding;
* Suspicion of intraductal extension or multifocality by mammography or MRI;
* Tumour not visible by ultrasound;
* Diameter > 2 cm;
* Distance to muscle or skin <1 cm;
* Lobular carcinoma;
* Intraductal carcinoma in > 20% of the biopsy sample
* Patients undergoing neoadjuvant chemotherapy or hormonotherapy.

Min Age: 40 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2013-09; Primary Completion 2017-07 (Actual); Study Completion 2017-07 (Actual)

PRIMARY OUTCOMES:
Intraoperative free margins (distance between the tumor and the margin in order to indicate if extensions are mandatory.) | 1 hour
  The pathologist performed a macroscopic study of the specimen, measuring the distance between the tumor and the margin in order to indicate if extensions are mandatory.

SECONDARY OUTCOMES:
Security of RFA (Adverse effects and cosmetic result) | 15 days
  Adverse effects and cosmetic result will be evaluated 15 days after the procedure
Efficacy of RFA (Tumoral viability in the ablation zone) | 7 days
  Tumoral viability in the ablation zone will be evaluated by NADH-diaphorase, COX and tunel

CONTACTS AND LOCATIONS:
Overall Officials: Amparo Garcia-Tejedor, MDPhD, Principal Investigator — Hospital Universitario Bellvitge-Idibell_Universidad de Barcelona
Locations (1):
- Hospital Universitario Bellvitge, L'Hospitalet de Llobregat, Barcelona, Spain

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Garcia-Tejedor A, Guma A, Soler T, Valdivieso A, Petit A, Contreras N, Chappuis CG, Falo C, Pernas S, Amselem A, Pla MJ, Fernandez-Montoli E, Burdio F, Ponce J. Radiofrequency Ablation Followed by Surgical Excision versus Lumpectomy for Early Stage Breast Cancer: A Randomized Phase II Clinical Trial. Radiology. 2018 Nov;289(2):317-324. doi: 10.1148/radiol.2018180235. Epub 2018 Aug 21. PMID 30129904